CLINICAL TRIAL: NCT05228951
Title: Pyrotinib Maleate, Trastuzumab, SHR6390(Dalpiciclib) and Letrozole in Combination for Neoadjuvant Treatment of Stage II-III TPBC
Brief Title: Pyrotinib Maleate, Trastuzumab, SHR6390 and Letrozole in Combination for Stage II-III TPBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Professor, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shengjing-LCG011
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; pyrotinib maleate; letrozole; SHR6390; trastuzumab; dalpiciclib
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; Trastuzumab; Letrozole; Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: single arm study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib maleate, dalpiciclib, Trastuzumab, letrozole (Experimental): After providing written informed consent, the participants will undergo combined treatment of pyrotinib maleate, CDK4/6 inhibitor dalpiciclib, trastuzumab and letrozole. The effectiveness of the combined treatment will be evaluated by MRI every two treatment cycles. If the disease progresses, the participant will withdraw from the trial. If the combined treatment has identified effectiveness, the participant will undergo surgical treatment within 4 weeks (over 2 weeks) after termination of the neoadjuvant treatment. The patients will be followed up for 5 years.
  Interventions: Drug: Pyrotinib maleate, dalpiciclib, Trastuzumab, letrozole

INTERVENTIONS:
Drug: Pyrotinib maleate, dalpiciclib, Trastuzumab, letrozole — After providing written informed consent, the participants will undergo combined treatment of pyrotinib maleate, CDK4/6 inhibitor dalpiciclib, trastuzumab and letrozole. The effectiveness of the combined treatment will be evaluated by MRI every two treatment cycles. If the disease progresses, the participant will withdraw from the trial. If the combined treatment has identified effectiveness, the participant will undergo surgical treatment within 4 weeks (over 2 weeks) after termination of the neoadjuvant treatment. The patients will be followed up for 5 years.
  Other Names: combined treatment

SUMMARY:
NOAH study confirmed that trastuzumab combined with chemotherapy can significantly improve PCR compared with chemotherapy alone, and established the status of trastuzumab as a new adjuvant targeted therapy. The emergence of CDK4/6 inhibitors has brought hope to breast cancer patients resistant to endocrine therapy. studies have shown that pyrotinib maleate combined with CDK4/6 inhibitor can significantly inhibit the proliferation of HER2 positive breast cancer cell lines, reduce the activation of pAKT and pHER3, inhibit cell arrest in G0-G1 phase, and increase cell apoptosis. In the mouse model, pyrotinib maleate combined with CDK4/6 inhibitor exhibits higher anti-tumor activity than any anti-tumor drug alone. Moreover, the toxicity of the combined therapy does not increase compared with monotherapy. This provides a good preclinical model for the treatment of breast cancer by pyrotinib maleate combined with CDK4/6 inhibitor.

In addition, NeoALTTO study、CALGB 40601 study、NSABP B-41 study confirmed that the clinical efficacy of lapatinib combined with trastuzumab combined chemotherapy was better than that of lapatinib or trastuzumab single target treatment group. Therefore, it is envisaged that the combination of pyrotinib maleate and dalpiciclib combined with letrozole on the basis of adding new trastuzumab to treat triple positive breast cancer will further improve the curative effect.

In conclusion, we believe that pyrotinib maleate combined with trastuzumab, dalpiciclib and letrozole can provide better strategies for neoadjuvant therapy in patients with II-III three positive breast cancer.

DETAILED DESCRIPTION:
This multi-center, single-arm, open-label trial will include 12 patients with stage II-III triple-positive breast cancer. After providing written informed consent, the participants will undergo combined treatment of pyrotinib maleate, CDK4/6 inhibitor dalpiciclib, trastuzumab，and letrozole. The effectiveness of the combined treatment will be evaluated by MRI every two treatment cycles. If the disease progresses, the participant will withdraw from the trial. If the combined treatment has identified effectiveness, the participant will undergo surgical treatment within 4 weeks (over 2 weeks) after termination of the five treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged≥18 years and ≤75 years meeting one of the following conditions;

   1. Those previously receiving ovariectomy, or aged ≥60 years
   2. Those aged < 60 years who have had 12 consecutive months of amenorrhoea without any pathological or physical causes, and have postmenopausal E2 and follicle stimulating hormone (FSH) levels
   3. Premenopausal or perimenopausal women who are willing to receive LHRH agonist treatment during the study period
2. Women who have breast cancer histopathologically confirmed by positive estrogen receptor (ER; >10%), positive progesterone receptor (PR; >1%), and positive human epidermal growth factor receptor 2 (HER2) according to the 2018 American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) human epidermal growth factor receptor 2 (HER2) guideline. ER, PR and HER2 will be assessed by immunohistochemistry (IHC) on harvested tissue. ER, PR and HER2 will be considered positive if the IHC result is positive (score 3+), or the IHC result is positive (2+) and in situ hybridization (ISH) amplification rate (≥2.0);
3. Women having stage II-III breast cancer diagnosed based on AJCC cancer staging system (8th edition) who will be admitted because of breast cancer for the first time;
4. Karnofsky Performance Status (KPS) Scale score ≥70;
5. The functional level of organs must meet the following requirements:

   a) Bone marrow function i) Absolute neutrophil count（ANC）≥1.5×109/L (no use of growth factor within 14 days) ii) Platelet count（PLT）≥100×109/L (no corrective treatment within 7 days) iii) Hemoglobin level（Hb）≥100 g/L (no corrective treatment within 7 days) b) Liver and kidney function i) Total bilirubin（TBIL）≤1.5 upper limit of normal value (ULN) ii) Alanine transaminase (ALT) and aspartate transaminase (AST) ≤3×ULN iii) Blood urea nitrogen (BUN) and creatinine ≤1.5×ULN and creatinine clearance≥50 mL/min (Cockcroft-Gault formula); c) Color Doppler echocardiography: Left ventricular ejection fraction ≥50% d) 12-lead electrocardiography: QTc interval ≤480 ms
6. Women who can undergo a biopsy;
7. Volunteers to participate in the study, provision of signed informed consent, good compliance and willingness to cooperate with follow-ups.

Exclusion Criteria:

1. Women who have received any form of anti-tumor treatment - (chemotherapy, radiotherapy, molecular targeted therapy, or endocrine therapy);
2. Those who have received other anti-tumor drug treatments concurrently;
3. Those who have bilateral breast cancer, inflammatory breast cancer or occult breast cancer;
4. Those who have stage IV breast cancer;
5. Those who have breast cancer not histopathologically confirmed;
6. Those who have other malignant tumors (with the exception of healed cervical carcinoma in situ) occurring in the past 5 years;
7. Those who have severe dysfunction of the heart, liver, kidney, and other major organs;
8. There are multiple factors that affect drug administration and absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
9. Those who have participated in other clinical drug trials in the past 4 weeks;
10. Those who are known to have a history of allergy to the component of study drugs; those who have a history of immunodeficiency, including positive detection of human immunodeficiency virus, hepatitis C virus, active hepatitis B or other acquired, congenital immunodeficiency diseases, or organ transplantation;
11. Those who had suffered from any heart disease, including arrhythmia which requires drug treatment or is of clinical significance; myocardial infarction; heart failure; and any other heart disease judged by the investigator as unsuitable for this trial;
12. Pregnant and lactating women; fertile women who provide positive results of baseline pregnancy test; women of childbearing age who are unwilling to take effective contraceptive measures during the whole study period;
13. If the accompanying diseases (including, but not limited to, severe hypertension, severe diabetes, and active infection, which cannot be controlled by drugs) that would be a potential hazard to participant's health, or affect the completion of the study as per investigator's judgement;
14. A clear history of neurological or psychiatric disorders, including epilepsy or dementia. Upon the suggestion of the investigators for other reasons

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (tpCR) | 1 month to 5 years after surgery
  tpCR is defined as the absence of residual invasive cancer on resected breast specimen and the sampled regional lymph nodes as shown by hematoxylin-eosin staining after completion of the neoadjuvant treatment

SECONDARY OUTCOMES:
Best overall response rate (BORR) | During neoadjuvant treatment(1-5 months of treatment)
  The proportion of patients who respond to the treatment at any study time point
Breast pathologic complete response (bpCR) | 1 month to 5 years after surgery
  There was no invasive carcinoma in the primary breast lesions (ypT0-is)
Residual cancer burden (RCB) | 1 month to 5 years after surgery
  RCB score is obtained according to pathological evaluation after completion of neoadjuvant treatment and surgery
Overall survival (OS) | Within 5 years after surgery
  It refers to the length of time from the start of treatment to the death of the patient
Disease-free survival (DFS) | Within 5 years after surgery
  It refers to the length of time from the start of medication after enrollment to the death of the patient because of the recurrence, distant metastasis of the disease, invasive contralateral breast cancer, or any other cause
Subject safety | From signing the informed consent to 28 days after last dose
  Number of Adverse Events using NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Cai-Gang Liu, PHD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will indicate whether pyrotinib maleate, CDK4/6 inhibitor SHR6390 and letrozole for treatment of stage II-III triple-positive breast cancer is safe and effective
Supporting Information: Study Protocol
Time Frame: 6 months to 5 years after publication
Access Criteria: Unlimited